CLINICAL TRIAL: NCT05741268
Title: Effect of Dialectical Behavior Therapy on Emotion Regulation Difficulties, Distress Tolerance, and Social Functioning Among Patients With Bipolar Disorder: A Randomized Controlled Trial
Brief Title: Effect of Dialectical Behavior in Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, assistant professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15122022
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-07

CONDITIONS: Dialectical Behavior Therapy
MeSH Terms: interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical behavior therapy (Experimental): Dialectical behavior therapy will be applied through psychoeducation, discussion, rehearsal, and homework assignments. Four modules were administered in Mindfulness, Emotion Regulation, Emotion Regulation, and Emotion Regulation.
  Interventions: Behavioral: Dialectical behavior therapy
- Routine psychological care (Active Comparator): they will receive psychological care such as stress management and social skills training.
  Interventions: Behavioral: Dialectical behavior therapy

INTERVENTIONS:
Behavioral: Dialectical behavior therapy — 14) Dialectical behavior therapy will be applied through psychoeducation, discussion, rehrasal and homework assignments. It contains four modules were administered in 14) Dialectical behavior therapy will be applied through psychoeducation, discussion, rehrasal and homework assignments. It contains four modules were administered in the following sequence 1. Mindfulness , 2. Emotion Regulation , 3. Distress Tolerance and 4. Interpersonal effectiveness.

SUMMARY:
This study aims to:

• Determine the effect of implementing Dialectical Behavior Therapy on emotion regulation difficulties, distress tolerance, and social functioning among patients with bipolar disorder.

RESEARCH HYPOTHESIS Patients with bipolar disorder who are exposed to Dialectical Behavior Therapy will exhibit lower emotion regulation difficulties, distress tolerance, and higher social functioning than those who are not exposed to such training.

DETAILED DESCRIPTION:
The researchers decided to work on a convenient sample of 30 adult patients with bipolar disorder. Dialectical behavior therapy will be applied through psychoeducation, discussion, rehearsal, and homework assignments. Four modules were administered in Mindfulness, Emotion Regulation, Emotion Regulation, and Emotion Regulation.

ELIGIBILITY:
Inclusion Criteria:1. Diagnosed with bipolar disorder for at least one month according to DSM V with no co-morbidity.

2. Their age does not exceed 60 years old. 3. Able to read and write. 4. Able & willing to participate in the study. 5. Living in Alexandria Governorate, Egypt.

Exclusion Criteria: demonstrate severe psychopathological symptom ( i.e: patient in acute stage)

-

Ages: 50 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotional Regulation Scale (DERS) | 2 weeks
  This tool (DERS) is a 36-items self-report scale developed by Gratz and Roemer (2004) to assess emotion regulation difficulties. The scale items are classified into six general subscales; non- acceptance of emotional responses (6 items); difficulty engaging in goal-directed behaviors (5 items); impulse control difficulties (6 items); lack of emotional awareness (6 items); limited access to emotional regulation strategies (8 items), and lack of emotional clarity (5 items).

SECONDARY OUTCOMES:
Distress Tolerance Scale (DTS) | 2 weeks
  The DTS (Simons & Gaher, 2005) is a 15-item selfreport questionnaire that assesses tolerance of distress, appraisal of distress, attention absorbed by negative emotions, and regulation efforts to alleviate distress. Items are rated on a 1 to 5 scale (1 = strongly agree; 5 = strongly disagree) with lower scores indicating poorer tolerance of distress. The DTS scale has demonstrated good test-retest reliability. In the current study the internal consistency of the DTS was excellent (Cronbach's α = .92).

OTHER OUTCOMES:
Social Functioning Scale (SFS) | 2 weeks
  The SFS is a 79-items self-report scale developed by Birchwood et al. (1990) to assess areas of social functioning of individuals with schizophrenia. The items are classified into seven subscales; withdrawal/social engagement (5 items), interpersonal communication (4 items), independence-performance (13 items), independence-competence (13 items), recreation (15 items), prosocial activities (22 items), and employment/occupational (5 items), in addition to two unscored preliminary questions (The latter two questions were excluded as they were measured in tool I).

CONTACTS AND LOCATIONS:
Overall Officials: Eman Taha, Study Chair — Egypt Faculty of Nursing Alexandria, Egypt
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Musket CW, Hansen NS, Welker KM, Gilbert KE, Gruber J. A pilot investigation of emotional regulation difficulties and mindfulness-based strategies in manic and remitted bipolar I disorder and major depressive disorder. Int J Bipolar Disord. 2021 Jan 4;9(1):2. doi: 10.1186/s40345-020-00206-0. PMID 33392824
- [Background] Miola A, Cattarinussi G, Antiga G, Caiolo S, Solmi M, Sambataro F. Difficulties in emotion regulation in bipolar disorder: A systematic review and meta-analysis. J Affect Disord. 2022 Apr 1;302:352-360. doi: 10.1016/j.jad.2022.01.102. Epub 2022 Jan 29. PMID 35093412
- [Background] Dodd AL, Gilbert K, Gruber J. Beliefs about the automaticity of positive mood regulation: examination of the BAMR-Positive Emotion Downregulation Scale in relation to emotion regulation strategies and mood symptoms. Cogn Emot. 2020 Mar;34(2):384-392. doi: 10.1080/02699931.2019.1626700. Epub 2019 Jun 7. PMID 31174453
- [Background] Eisner L, Eddie D, Harley R, Jacobo M, Nierenberg AA, Deckersbach T. Dialectical Behavior Therapy Group Skills Training for Bipolar Disorder. Behav Ther. 2017 Jul;48(4):557-566. doi: 10.1016/j.beth.2016.12.006. Epub 2017 Jan 6. PMID 28577590